CLINICAL TRIAL: NCT04304391
Title: The Determination of the Operative Temperature Levels Using Er:YAG Laser and Diode Laser Supported Resective Gingival Surgery and the Clinical and Biochemical Evaluation of it's Effect on Postoperative Imflammation, Epithelization and Pain
Brief Title: Evaluation of Healing Process After Laser Asissted Gingivectomy Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, mehmet murat taskan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TOGUGKARA
Record Dates: First submitted 2020-03-06; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Gingival Enlargement
MeSH Terms: conditions — Gingival Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): Conventional Gingivectomy:Technique is performed with conventional surgical instruments.
  Interventions: Procedure: Resective Gingival Surgery
- Group B (Experimental): Diode Laser Assisted Gingivectomy: Technique is performed with using diode laser.
  Interventions: Procedure: Resective Gingival Surgery
- Group C (Experimental): Er:YAG Laser Assisted Gingivectomy: Technique is performed with using Er:YAG laser.
  Interventions: Procedure: Resective Gingival Surgery
- Group D (No Intervention): Negative Control Group

INTERVENTIONS:
Procedure: Resective Gingival Surgery — Gingivectomy and gingivoplasty:Resective gingival surgical procedured
  Arms: Group A; Group B; Group C

SUMMARY:
Objective: The aim of this study was to evaluate and determine clinical and biochemical comparison of 3 different methods including Er:YAG laser, diod laser, and conventional techniques.

Method: This study was conducted on 32 female, 13 male, a total of 45 individuals (study group patients) with an indication of resective gingival surgery in the anterior region of the maxillar anterior regions and 11 female, 4 men, a total of 15 individuals (negative control group patients) with a healthy gingiva. Clinical periodontal parameters, gingival crevicular fluid (GCF) KGF-2 and VEGF-A levels and gingival temperature levels were recorded before the investigation and during operations with 3 different techniques, gingival temperature was measured. Gingival temperature and epithelization levels in 3, 7, 14 and 21 days; GCF KGF-2 and VEGF-A levels in 14 and 21 days and pain levels between 1-7 days of post-operative healing process were evaluated. Preoperative anxiety and postoperative satisfaction were evaluated through questionnaires

DETAILED DESCRIPTION:
Objective: The aim of this study was to evaluate and determine clinical and biochemical comparison of 3 different methods including Er:YAG laser, diod laser, and conventional techniques commonly used in resective gingival surgeries in terms of preoperative anxiety, postoperative satisfaction, epithelization, gingival temperature, inflammation and pain levels in post-operative healing process.

Method: This study was conducted on 32 female, 13 male, a total of 45 individuals (study group patients) with an indication of resective gingival surgery in the anterior region of the maxillar anterior regions and 11 female, 4 men, a total of 15 individuals (negative control group patients) with a healthy gingiva. Clinical periodontal parameters, gingival crevicular fluid (GCF) KGF-2 and VEGF-A levels and gingival temperature levels were recorded before the investigation and during operations with 3 different techniques, gingival temperature was measured. Gingival temperature and epithelization levels in 3, 7, 14 and 21 days; GCF KGF-2 and VEGF-A levels in 14 and 21 days and pain levels between 1-7 days of post-operative healing process were evaluated. Preoperative anxiety and postoperative satisfaction were evaluated through questionnaires

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy individuals
* the existence of at least 20 functioning teeth,
* the existence of chronic inflammatory gingival enlargement

Exclusion Criteria:

* pregnancy/lactation,
* drug use,
* previous periodontal therapy within 6 months

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of Gingival Temperature | 6 months
  Operative and post operative gingival temperature levels of the application region measured and recorded with using a noncontact infrared thermometer. The temperature measurement during the process was performed by an infrared thermometer (Optris GMBH, Manuel LS, Berlin, Germany). The device had a measurement and recording range from -35 ° C to 900 ° C, optical resolution 75: 1, thermal resolution 0.1 ° C, waveband range 8-14, USB interface and graphical software program.
Evaluation of Gingival Epithelization | 6 months
  Epithelization levels of resection region were measured and evaluated with using Image J software. Wound surface epithelization in the healing process was evaluated with a staining solution (Mira-2-tone, GMBH & Co., Duisburg, Germany). The treatment area was isolated. The solution carrier was applied with cotton pellets. The excess solution was removed by air-water spray. The standardized photographs were taken and transferred to the java based analysis program (Image J 1.31o, National Institutes of Health, Bethesda, MD, USA). The dark stained areas were calculated in the computer environment

SECONDARY OUTCOMES:
Evaluation of Gingival Pain Levels: Visual Analog Scale | 6 months
  Pain levels were evaluated with Visual Analog Scale in post operative process.A visual analogue scale (VAS) was used to evaluate pain after surgeries. Patients were asked to mark the pain levels at the levels from 0 (no pain) to 10 (the most severe pain) on the scale

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided